CLINICAL TRIAL: NCT05662618
Title: Prospective, Multicenter, Randomized Controlled Clinical Trial to Verify the Efficacy and Safety of Rapamycin Coated Peripheral Balloon Catheter in the Treatment of Femoral Popliteal Artery Disease
Brief Title: To Verify the Efficacy and Safety of Rapamycin Coated Peripheral Balloon Catheter in the Treatment of Femoral Popliteal Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Bomaian Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LFBMA-202201
Record Dates: First submitted 2022-12-01; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapamycin coated peripheral balloon catheter (Experimental): Rapamycin coated peripheral balloon catheter of Bomaian Company.
  Interventions: Procedure: Percutaneous selective arteriography of peripheral arteries
- Drug eluting peripheral balloon catheter (Active Comparator): Paclitaxel eluting balloon catheter
  Interventions: Procedure: Percutaneous selective arteriography of peripheral arteries

INTERVENTIONS:
Procedure: Percutaneous selective arteriography of peripheral arteries — Treatment of stenosis or occlusion of superficial femoral artery and/or popliteal artery with rapamycin coated balloon catheter.
Procedure: Percutaneous selective arteriography of peripheral arteries — Paclitaxel coated balloon catheter for the treatment of stenosis or occlusion of superficial femoral artery and/or popliteal artery.

SUMMARY:
A prospective randomized trial to validate the efficacy and safety of rapamycin coated peripheral balloon catheter in the treatment of femoral popliteal artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with arteriosclerosis obliterans of lower extremities, and Rutherford's rating is 2-5.
* Patients with severe stenosis (≥ 70%) or occlusion of superficial femoral artery and/or proximal popliteal artery (within P1 stage)
* Patients with total length of target lesion ≤ 20cm and length of occluded segment ≤ 15cm (the distance between two segments of lesions less than 2cm is considered as the same lesion)
* Those who agree to participate in this clinical trial and sign the informed consent form Exclusion criteria：
* This operation is planned to intervene patients with bilateral lower limbs.
* Patients whose guide wire fails to pass through the target lesion.
* Patients whose target lesion is in stent restenosis (ISR).
* ≥ 2 lesions need to be treated in the target vessel (if the distance between two lesions is less than 2cm, it is considered as the same lesion).
* Patients with target lesions requiring rotary resection/laser therapy/thrombus aspiration for this treatment.
* Patients with ipsilateral iliac artery inflow tract lesions that cannot be successfully treated (i.e. residual stenosis ≥ 30% after treatment).
* There is less than one unobstructed blood vessel under the knee of the target limb before operation (unobstructed is defined as visual stenosis<50%).
* Residual stenosis ≥ 30% after pre expansion of target lesion or severe (≥ Grade D) flow limiting dissection.
* Patients with obviously abnormal renal function (creatinine > 2.5mg/dL or 220umol/L) or undergoing dialysis.
* Patients with severe liver dysfunction who are judged by the researcher to be unsuitable for surgery.
* Patients with severe coagulation dysfunction or uncontrolled severe infection who are not suitable for surgery.
* Patients who have performed distal amputation (above metatarsal) on the affected or opposite limb in the past.
* Patients who received local or systemic thrombolytic therapy within 48 hours before surgery.
* Patients receiving vascular interventional therapy or surgical treatment on target limb within 30 days before operation.
* Patients known to be allergic to aspirin, clopidogrel, paclitaxel and rapamycin.
* Pregnant or lactating women and patients with family planning during the study
* Patients who are participating in clinical trials of other drugs or medical devices but are not included in the group.
* Patients with life expectancy less than 12 months
* Patients not suitable for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2022-12-31 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
primary patency rate, PPR. | 12months
  It is defined as:Primary patency of target lesion: the target lesion is patency (systolic peak blood flow ratio<2.4) and there is no clinically driven target lesion revascularization (TLR) by Doppler ultrasound.

SECONDARY OUTCOMES:
Device success rate | The day of operation.
  It is defined as: the balloon catheter can reach the target lesion, expand successfully, without rupture, and withdraw successfully.
Operation success rate | 1DAY
  The success of surgery was defined as: residual stenosis ≤ 50% (without salvage stent implantation) or ≤ 30% (with salvage stent implantation).
Target Lesion Revascularization incidence. | 12 months after operation.
  Target Lesion Revascularization is defined as any re intervention treatment required in the target lesion.

OTHER OUTCOMES:
Incidence rate of major adverse events | 12 months after operation.
  Major adverse events were defined as: all cause death at 30 days, amputation of diseased limbs 12 months after operation, and clinically driven target vessel revascularization
Occurrence of other adverse events and serious adverse events | 12 months after operation.
  Evaluation method: other adverse events and serious adverse events of the subjects were recorded through telephone/hospital visit.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Medical Center of the General Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No